CLINICAL TRIAL: NCT01870466
Title: A Randomized, Open-label, Multiple-dose, Crossover Study to Investigate the Pharmacodynamic Drug Interaction Between Cilostazol and Statins in Healthy Male Volunteer
Brief Title: Pharmacodynamic Drug Interaction Between Cilostazol and Statins
Acronym: SMCCPT-100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-11-004
Record Dates: First submitted 2012-05-04; First posted 2013-06-06 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
MeSH Terms: interventions — Cilostazol; Simvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- C -> C + S (Experimental): cilostazol (C) in period 1, cilostazol + simvastatin (C+S) in period 2
  Interventions: Drug: Cilostazol; Drug: Simvastatin
- C + S -> C (Experimental): cilostazol + simvastatin (C+S) in period 1, cilostazol (C) in period 2
  Interventions: Drug: Cilostazol; Drug: Simvastatin
- S -> S + C (Experimental): simvastatin (S) in period 1, simvastatin + cilostazol (S+C) in period 2
  Interventions: Drug: Cilostazol; Drug: Simvastatin
- C + S -> S (Experimental): cilostazol + simvastatin (C+S) in period 1, simvastatin (S) in period 2
  Interventions: Drug: Cilostazol; Drug: Simvastatin
- R -> C + R (Experimental): rosuvastatin (R) in period 1, cilostazol + rosuvastatin (C+R) in period 2
  Interventions: Drug: Cilostazol; Drug: Rosuvastatin
- C + R -> R (Experimental): cilostazol + rosuvastatin (C+R) in period 1, rosuvastatin (R) in period 2
  Interventions: Drug: Cilostazol; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Cilostazol — cilostazol bid for 7 days
  Other Names: cilostazol (C); Plettal 100 mg
Drug: Simvastatin — simvastatin qd for 7 days
  Other Names: simvastatin (S); Zocor 40 mg
  Arms: C + S -> C; C + S -> S; C -> C + S; S -> S + C
Drug: Rosuvastatin — rosuvastatin qd for 7 days
  Other Names: Rosuvastatin (R); Crestor 20 mg
  Arms: C + R -> R; R -> C + R

SUMMARY:
The purpose of this study is to evaluate pharmacodynamic drug interaction between cilostazol and statins (simvastatin as a CYP3A substrate and rosuvastatin as a non-CYP3A substrate) in healthy male subjects.

DETAILED DESCRIPTION:
Subjects suitable for this study will visit to the Clinical Trial Center, Samsung Medical Center for 7 days and pharmacodynamic samplings will be performed following the administration of study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20 - 55 years
* A body mass index in the range 18.5 - 27 kg/m2
* Willingness to participate during the entire study period
* Written informed consent after being fully informed about the study procedures

Exclusion Criteria:

* Any past medical history of hepatic, renal, neurologic, cardiovascular, respiratory, endocrine, hemato-oncologic or psychiatric disease
* Active bleeding or bleeding tendency
* History of gastrointestinal disease or surgery possibly affecting drug absorption
* History of clinically significant drug hypersensitivity
* Use of medication within 7 days before the first dose
* Heavy drinker (>140 g/week)
* Whole blood donation during 60 days before the study
* Judged not eligible for study participation by investigator

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
lipid lowering effect | 7 days
  lipid panel

SECONDARY OUTCOMES:
anti-platelet effect | 7 days
  platelet aggregation test

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Wook Ko, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea